CLINICAL TRIAL: NCT02834338
Title: Usage of Activity Tracking in Major Visceral Surgery - the Enhanced Perioperative Mobilization (EPM) Trial
Brief Title: Enhanced Perioperative Mobilization (EPM) Trial
Acronym: EPMIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TW-003
Record Dates: First submitted 2016-06-15; First posted 2016-07-15 (Estimated); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Pancreatic Resection; Liver Resection; Gastric Resection; Colorectal Resection
Keywords: activity tracking; postoperative recovery; ERAS; fast-track surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Laparoscopic surgery, control (No Intervention): The control group is wearing an activity tracker wristband with covered display, so that the step count can't be read out.
- Laparoscopic surgery, intervention (Active Comparator): activity tracking for autofeedback
  Interventions: Device: activity tracking for autofeedback
- Open surgery, control (No Intervention): The control group is wearing an activity tracker wristband with covered display, so that the step count can't be read out.
- Open surgery, intervention (Active Comparator): activity tracking for autofeedback
  Interventions: Device: activity tracking for autofeedback

INTERVENTIONS:
Device: activity tracking for autofeedback — The intervention group receives an unblinded wristband. The handling of the activity trackers is explained to the patients and a predefined mobilization end-point (step-count) for the first five PODs is targeted. The target step-count was set at the 85% quartile obtained from a previous pilot study. The patients are assessed and monitored two times daily between 9 and 11 o'clock AM and between 3 and 5 o'clock PM by a surgical fellow or a study nurse throughout their hospital stay for read-out of the step count, assurance of the proper use and functioning, and for communication of the autofeedback.
  Arms: Laparoscopic surgery, intervention; Open surgery, intervention

SUMMARY:
Randomized Controlled Trial to monitor and increase the postoperative mobilization of the patients undergoing major visceral surgery by giving a continuous autofeedback of the step count using activity tracking wristbands.

DETAILED DESCRIPTION:
Patients undergoing elective open and laparoscopic surgery of colon, rectum, stomach, pancreas and liver for any indication will be included. Further inclusion criteria are: age between 18-75 years, ASA score < 4, and a signed informed consent. Patients are stratified into two subgroups (laparoscopic and open surgery) and will be randomized 1:1 for an autofeedback of their step-count using an activity tracker wristband or for the control group without autofeedback. Sample size (n = 29 patients in each of the four groups, overall n = 119) is calculated on an assumed difference in step-count of 250 steps daily (intervention versus control group). The primary study endpoint is the step-count during the first five postoperative days; secondary endpoints are the percentage of patients in the two groups, who master the predefined mobilization (step-count) targets, the assessment of additional activity data from the devices, the assessment of the preoperative mobility, length of hospital and intensive care unit stay, number of patients who receive physiotherapy, 30-day mortality, and the overall 30-day morbidity.

ELIGIBILITY:
Inclusion Criteria:

* elective laparoscopic and open surgery of the colon and rectum (colectomy, hemicolectomy, segment resection, rectum extirpation, deep anterior rectum resection, sigmoid resection, proctocolectomy), of the stomach (total, subtotal and atypical gastric resections), of the pancreas (any kind of pancreatic resections), and of the liver (hemihepatectomy, atypical resection, anatomical segment resection)
* ASA score < IV
* completed informed consent.

Exclusion Criteria:

* emergency surgery
* mental inability to complete postoperative assessment protocols
* preoperatively immobile patients

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
Median Step count | First to fifth postoperative day

SECONDARY OUTCOMES:
Percentage of patients, who master the predefined mobilization (step-count) targets | First to fifth postoperative day
Distance (km) | First to fifth postoperative day
  Assessed by the activity tracker wristband
Activity time (min.) | First to fifth postoperative day
  Assessed by the activity tracker wristband
inactivity | First to fifth postoperative day
  Assessed by the activity tracker wristband
calorie consumption (kcal) | First to fifth postoperative day
  Assessed by the activity tracker wristband
Compliance | First to fifth postoperative day
  Compliance to wear the wrist band
Assessment of the preoperative mobility | Preoperative
  Measured by International Physical Activity Questionnaire (IPAQ)
Length of hospital stay | 30 days
Length of ICU stay | 30 days
Amount of patients which receive physiotherapy | First to fifth postoperative day
Mortality | 30 days
Overall morbidity | 30 days
  According the Clavien-Dindo classification

CONTACTS AND LOCATIONS:
Overall Officials: Thilo Welsch, MD, MBA, Principal Investigator — Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, Technical University of Dresden, Germany
Locations (1):
- Department of Visceral, Thoracic and Vascular Surgery, University Hospital Carl Gustav Carus, Technical University of Dresden, Dresden, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wolk S, Linke S, Bogner A, Sturm D, Meissner T, Mussle B, Rahbari NN, Distler M, Weitz J, Welsch T. Use of Activity Tracking in Major Visceral Surgery-the Enhanced Perioperative Mobilization Trial: a Randomized Controlled Trial. J Gastrointest Surg. 2019 Jun;23(6):1218-1226. doi: 10.1007/s11605-018-3998-0. Epub 2018 Oct 8. PMID 30298422
- [Derived] Wolk S, Meissner T, Linke S, Mussle B, Wierick A, Bogner A, Sturm D, Rahbari NN, Distler M, Weitz J, Welsch T. Use of activity tracking in major visceral surgery-the Enhanced Perioperative Mobilization (EPM) trial: study protocol for a randomized controlled trial. Trials. 2017 Feb 21;18(1):77. doi: 10.1186/s13063-017-1782-1. PMID 28222805